CLINICAL TRIAL: NCT06935305
Title: One Step Nucleic Acid Amplification (OSNA) Versus Ultrastaging to Detect Sentinel Lymph Node Metastasis in Endometrial Cancer: a Randomized, Multicenter, Controlled Trial (SENT-OSNA Study)
Brief Title: OSNA Versus Ultrastaging to Detect Sentinel Lymph Node Metastasis in Endometrial Cancer
Acronym: SENT-OSNA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Sysmex Europe GmbH (Industry)
Responsible Party: Principal Investigator, Fanfani Francesco, Professor Francesco Fanfani, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7170
Record Dates: First submitted 2025-02-09; First posted 2025-04-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; OSNA; sentinel lymph node; ultrastaging
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized before surgery: in one study arm, the search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the ultrastaging method (standard), while in the other arm it will be conducted using the OSNA method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrastaging arm (Active Comparator): In this study arm, the search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the ultrastaging method (standard)
  Interventions: Device: Ultrastaging
- OSNA arm (Experimental): In this arm the search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the OSNA method (experimental)
  Interventions: Device: OSNA

INTERVENTIONS:
Device: OSNA — The search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the OSNA method
  Arms: OSNA arm
Device: Ultrastaging — The search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the ultrastaging method
  Arms: ultrastaging arm

SUMMARY:
Patients enrolled in the study will be randomized before surgery: in one study arm, the search for lymph node metastases in surgically removed sentinel lymph nodes will occur using the ultrastaging method (standard), while in the other arm it will be conducted using the OSNA method.

DETAILED DESCRIPTION:
This is a non-inferiority randomized trial with the incidence of patients with metastatic SLN as primary endpoint. Based on recent literature, incidence of patients with metastatic SLN detected by ultrastaging has an average value of 11%. Assuming a -4% as the maximum allowable difference in detection rate to declare non-inferiority, a power of 80% and a significance level of 2.5% (one-side) a sample size of 1922 (961 per arm) is needed. Two interim analyses are planned, one after the first 640 and the second after 1280 patients. At the first interim analysis null hypothesis (inferiority of OSNA with respect to ultrastaging) will be rejected at a significance level <0.00010 otherwise the study will go on and at the second analysis the null hypothesis will be rejected at a significance level of 0.0059. The final analysis will use 0.0189 as significance threshold. The O'Brien Fleming alpha spending function was used to define these values.

The primary endpoint is defined as the proportion of patients with positive SLN over the total of randomized patients. This proportion will be reported together with the 95% confidence interval to better identify the range of inferential values. Incidence of isolated tumor cells, micro- and macro-metastasis will be calculated.

Number of copies of CK19 mRNA to define volume of metastases will be adapted from previous reports.

To describe the sample, quantitative variables will be summarized using median and interquartile range while categorical items will be reported as absolute counts and percentages. Patients will be described according the arm they were randomized to. A first analysis will be performed on an Intent-To-Treat basis, considering all randomized patients. A secondary analysis will be performed on the Per-Protocol population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer
* Apparent (pre-operative) FIGO stage I-II
* Radical surgery
* Attempt of SLN mapping

Exclusion Criteria:

* Uterine sarcoma (including endometrial stromal sarcoma)
* Fertility sparing surgery
* Dedifferentiated histology
* Undifferentiated histology
* Neoadjuvant therapy
* Previous surgery to pelvic lymph nodes
* Lymph nodes with short axis >15 mm at pre-operative imaging

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1922 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2029-03-17 (Estimated)

PRIMARY OUTCOMES:
Number of SLN metastasis detected by OSNA versus ultrastaging method | From enrollment to the acquisition of the histological examination (8 weeks)
  We will evaluate the number of lymph node metastases identified with both methods, in order to calculate the incidence of lymph node metastases for each group

SECONDARY OUTCOMES:
Overall survival (measured in months) in patients with a diagnosis of lymph node metastases (identified with OSNA and ultrastaging), performing stratification by molecular class. | 3 years (a 3-year follow-up is planned)
  The aim is to assess the impact of both techniques on staging, prognosis, and therapeutic strategies, optimizing patient management according to molecular subtypes.
Disease-free survival (measured in months) in patients with a diagnosis of lymph node metastases (identified with OSNA and ultrastaging), performing stratification by molecular class. | 3 years (a 3-year follow-up is planned)
  The aim is to assess the impact of both techniques on staging, prognosis, and therapeutic strategies, optimizing patient management according to molecular subtypes.
3 year disease-free survival (measured in months) in OSNA versus ultrastaging negative patients | 3 years (a 3-year follow-up is planned)
  The study evaluates 3 year disease-free survival in endometrial carcinoma patients with negative sentinel lymph nodes (SLN) according to OSNA and ultrastaging. By comparing both techniques, the research aims to determine their prognostic value and potential implications for tailoring post-surgical management and follow-up strategies
3 year overall survival (measured in months) in OSNA versus ultrastaging negative patients | 3 years (a 3-year follow-up is planned)
  The study evaluates 3 year overall survival in endometrial carcinoma patients with negative sentinel lymph nodes (SLN) according to OSNA and ultrastaging. By comparing both techniques, the research aims to determine their prognostic value and potential implications for tailoring post-surgical management and follow-up strategies
5-year disease-free survival (measured in months) in OSNA versus ultrastaging negative patients | 5 years
  The study evaluates 5-year disease-free survival in endometrial carcinoma patients with negative sentinel lymph nodes (SLN) according to OSNA and ultrastaging. By comparing both techniques, the research aims to determine their prognostic value and potential implications for tailoring post-surgical management and follow-up strategies
5-year overall survival (measured in months) in OSNA versus ultrastaging negative patients | 5 years
  The study evaluates 5-year overall survival in endometrial carcinoma patients with negative sentinel lymph nodes (SLN) according to OSNA and ultrastaging. By comparing both techniques, the research aims to determine their prognostic value and potential implications for tailoring post-surgical management and follow-up strategies
Incidence of endosalpingiosis in ultrastaging arm | From enrollment to the acquisition of the histological examination (8 weeks)
  The study investigates the incidence of endosalpingiosis in the ultrastaging arm of sentinel lymph node analysis in endometrial carcinoma. The aim is to assess its frequency, potential clinical significance, and implications for pathological interpretation and patient management.
Total Tumor Load (calculating by summing the number of copies of CK19 from each sentinel lymph node) and correlation with prognosis | 3 years (a 3-year follow-up is planned)
  The study examines the total tumor load (TTL), defined as the sum of CK19 copies from each sentinel lymph node (SLN), and its correlation with prognosis.
Dimension of SLN (measured in millimeters) metastases at ultrastaging and correlation with prognosis | 3 years (a 3-year follow-up is planned)
  The study analyzes the size of sentinel lymph node (SLN) metastases detected through ultrastaging and its correlation with prognosis in endometrial carcinoma. The objective is to evaluate the prognostic significance of metastasis dimensions and their potential impact on clinical management and treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fanfani, Professor, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy, Italy

REFERENCES:
- [Background] Marchocki Z, Cusimano MC, Clarfield L, Kim SR, Fazelzad R, Espin-Garcia O, Bouchard-Fortier G, Rossi EC, Stewart KI, Soliman PT, How JA, Gotlieb WH, Holloway RW, Ianieri MM, Cabrera S, Lim YK, Ferguson SE. Sentinel lymph node biopsy in high-grade endometrial cancer: a systematic review and meta-analysis of performance characteristics. Am J Obstet Gynecol. 2021 Oct;225(4):367.e1-367.e39. doi: 10.1016/j.ajog.2021.05.034. Epub 2021 May 29. PMID 34058168
- [Background] Persson J, Salehi S, Bollino M, Lonnerfors C, Falconer H, Geppert B. Pelvic Sentinel lymph node detection in High-Risk Endometrial Cancer (SHREC-trial)-the final step towards a paradigm shift in surgical staging. Eur J Cancer. 2019 Jul;116:77-85. doi: 10.1016/j.ejca.2019.04.025. Epub 2019 Jun 7. PMID 31181536
- [Background] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, George S, Han E, Higgins S, Huh WK, Lurain JR 3rd, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Uterine Neoplasms, Version 1.2018, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2018 Feb;16(2):170-199. doi: 10.6004/jnccn.2018.0006. PMID 29439178
- [Background] Bodurtha Smith AJ, Fader AN, Tanner EJ. Sentinel lymph node assessment in endometrial cancer: a systematic review and meta-analysis. Am J Obstet Gynecol. 2017 May;216(5):459-476.e10. doi: 10.1016/j.ajog.2016.11.1033. Epub 2016 Nov 18. PMID 27871836
- [Background] Bogani G, Murgia F, Ditto A, Raspagliesi F. Sentinel node mapping vs. lymphadenectomy in endometrial cancer: A systematic review and meta-analysis. Gynecol Oncol. 2019 Jun;153(3):676-683. doi: 10.1016/j.ygyno.2019.03.254. Epub 2019 Apr 2. PMID 30952370
- [Background] Concin N, Matias-Guiu X, Vergote I, Cibula D, Mirza MR, Marnitz S, Ledermann J, Bosse T, Chargari C, Fagotti A, Fotopoulou C, Gonzalez Martin A, Lax S, Lorusso D, Marth C, Morice P, Nout RA, O'Donnell D, Querleu D, Raspollini MR, Sehouli J, Sturdza A, Taylor A, Westermann A, Wimberger P, Colombo N, Planchamp F, Creutzberg CL. ESGO/ESTRO/ESP guidelines for the management of patients with endometrial carcinoma. Int J Gynecol Cancer. 2021 Jan;31(1):12-39. doi: 10.1136/ijgc-2020-002230. Epub 2020 Dec 18. PMID 33397713
- [Background] Lortet-Tieulent J, Ferlay J, Bray F, Jemal A. International Patterns and Trends in Endometrial Cancer Incidence, 1978-2013. J Natl Cancer Inst. 2018 Apr 1;110(4):354-361. doi: 10.1093/jnci/djx214. PMID 29045681
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06935305/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06935305/ICF_001.pdf